CLINICAL TRIAL: NCT05220280
Title: Long-term Follow-up of a Randomized Multicenter Trial on Impact of Imatinib and Infliximab on Long-COVID in Hospitalized COVID-19 Patients
Brief Title: SOLIDARITY Finland Plus Long-COVID
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Clinical Urology and Epidemiology Working Group (Other Government)
Collaborators: University of Helsinki (Other); World Health Organization (Other); Helsinki University Central Hospital (Other); Hyvinkää Hospital (Other); Kanta-Häme Central Hospital (Other Government); Kuopio University Hospital (Other); City of Helsinki (Other); Oulu University Hospital (Other); Porvoo Hospital (Unknown); Seinajoki Central Hospital (Other); Mikkeli Central Hospital (Other); Tampere University Hospital (Other)
Responsible Party: Principal Investigator, Kari Tikkinen, Professor, University of Helsinki
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SOLP21
Record Dates: First submitted 2022-02-01; First posted 2022-02-02 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Coronavirus Disease 2019; SARS-CoV-2 Acute Respiratory Disease
Keywords: Long COVID; imatinib; infliximab
MeSH Terms: conditions — COVID-19; Post-Acute COVID-19 Syndrome | interventions — Imatinib Mesylate; Infliximab

STUDY DESIGN:
Masking Description: Open label trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Local standard of care (No Intervention)
- Imatinib + local standard of care (Experimental)
  Interventions: Drug: Imatinib
- Infliximab + local standard of care (Experimental)
  Interventions: Drug: Infliximab

INTERVENTIONS:
Drug: Imatinib — Oral imatinib 400 mg tablet once a day for 14 days.
  Arms: Imatinib + local standard of care
Drug: Infliximab — Infliximab is administered as a single IV infusion with the proposed dosing schedule of 5 mg/kg body weight.
  Arms: Infliximab + local standard of care

SUMMARY:
The SOLIDARITY PLUS Finland Long-COVID trial aims to assess the long-term effects of imatinib and infliximab, used during acute hospitalization due to COVID-19-infection, on long-COVID symptoms and quality of life (QoL) using questionnaires at six months, one and two years post-discharge. The primary research questions are whether imatinib or infliximab lower the risk of long-COVID symptoms and leads to better QoL in the long term.

Objectives include:

i) Long-COVID symptoms

To investigate the effect of imatinib (vs. usual care only) and infliximab (vs. usual care only) on the occurrence of symptoms that have been associated with the long-COVID syndrome. The questionnaires will take place at six months, one and two years after the hospital admission. The questionnaire will be the same that has been used in the SOLIDARITY Finland Long-COVID trial on remdesivir. The questionnaire was developed by our multidisciplinary team of physicians, including the representation of multiple specialties such as general practice, lung diseases, neurology, internal medicine, rheumatology, genetics, and clinical epidemiology, and two patient partners.

The symptom questionnaire - that will be completed by patients at one and two years - measures basic patient information (age, height, weight, smoking status, major comorbidity, and working status) and a wide variety of potential long-COVID-symptoms and their bother (1. Fatigue; 2. Attention deficits; 3. Memory problems; 4. Sleeping difficulties; 5. Depressive mood; 6. Anxiety; 7. Dizziness; 8. Headache; 9. Tinnitus; 10. Paresthesias; 11. Changes in taste/smell perceptions; 12. Postexertional malaise; 13. Palpitations; 14. Chest discomfort; 15. Nausea; 16. Skin rash; 17. Joint aches; 18. Muscle pains; 19. Continuous cough; 20. Respiratory tract mucous discharges).

ii) Quality of life

The EQ-5D-5L questionnaire will be used to compare patients' quality of life in imatinib, infliximab, and usual care arms.

EQ-5D-5L questionnaire assesses the following domains: 1. Mobility; 2. Self-care; 3. Usual activities; 4. Pain and discomfort; 5. Anxiety and depression; 6. The visual analog scale of subjective perception of overall health.

Additionally (at 1 or 2 years; depending on future funding and ethical approval decisions):

* The Finnish healthcare registries (such as Statistics Finland Mortality Database, the HILMO Care Register for Health Care, and/or Digital and Population Data Services Agency (Finnish Digital Agency)) will be used to estimate long-term mortality and incidence of major comorbidity in treatment arms.
* Lung function will be assessed using spirometry and diffusing capacity, as well as the six-minute walk test (6 mwt) in treatment arms.
* Whole-genome genotyping will be performed for a genome-wide association study to investigate genetic correlates of long-COVID-19 -symptoms in treatment arms.

DETAILED DESCRIPTION:
The SOLIDARITY Finland Plus Long-COVID is the long-term follow-up of the SOLIDARITY Finland Plus trial. With local adjustments, this clinical trial follows the WHO core protocol. SOLIDARITY Finland (Plus) is an adaptive, randomized, open-label clinical trial evaluating the safety and efficacy of imatinib, infliximab, and local standard of care in hospitalized adult patients diagnosed with COVID-19.)

Study population:

The study population consists of adult patients (18 years and older) with laboratory-confirmed SARS-2-CoV-2, who are admitted to the hospital ward or the intensive care unit (ICU). Adult hospital patients, with definite COVID-19 and, as per the responsible doctor, no contraindication to the study drugs were entered into the online electronic data collection system and randomly allocated (1:1:1, if no contraindications) between:

1. the local standard of care alone or
2. local standard of care plus oral imatinib (until discharge or up to 14 days) or
3. local standard of care plus a single intravenous infusion of infliximab.

Exclusion criteria:

There are several drug-specific exclusion criteria. Contraindications to be randomized to the infliximab study arm include tuberculosis, hepatitis B, severe bacterial infection, unstable cardiac insufficiency, multiple sclerosis, or hypersensitivity to infliximab, or previous regular use of biological medication with immunomodulatory effects. Contraindications to be randomized to imatinib include hepatitis B, liver cirrhosis, and hypersensitivity to imatinib.

In addition to drug-specific exclusion criteria, the trial also has several general exclusion criteria. These include very poor prognosis due to comorbidity ( an estimated less than three months life expectancy), ASAT/ALAT-ratio over five-fold the upper limit, severe renal failure (GFR < 30), acute myocardial infarction or unstable angina pectoris, pregnancy or breastfeeding.

Hospitalized patients are recruited from August 2021 onwards in participating hospitals to the SOLIDARITY Finland Plus trial. During patient recruitment and before randomization, the following data are to be collected (via the WHO database):

1. hospital and randomizing doctor
2. confirmation that patient has provided consent
3. patient identifiers, age, and sex
4. major comorbidities, including diabetes, heart disease, chronic lung disease, chronic liver disease, asthma, HIV infection, obesity
5. hospitalization date
6. COVID severity by

   1. possible respiratory support: no oxygen, low-flow oxygen, high-flow nasal oxygen, non-invasive ventilation, invasive ventilation, and ECMO.
   2. SpO2 (%) and respiratory rate.
7. Imaging abnormalities.
8. Locally available study drugs.

Consent:

All prospective patients for the long-term follow-up have already consented to SOLIDARITY Finland Plus during their hospital stay. In the SOLIDARITY Finland Plus Long-COVID, patients will receive, by mail, an information letter, consent form, and questionnaires. The mail will be sent three days before the three follow-up time points, which are at six months, one, and two years. Patients may reply by i) sending back the completed documents, ii) scheduling a phone call with an investigator for an interview, or iii) declining participation. If the patient does not reply in 21 days (from the day the investigators sent the questionnaire to the patient), the investigators will send one reminder by mail and, if there will not be a reply, then the investigators will approach the patient via telephone at around 14 (12-15) days from the reminder mail. The phone call will be attempted twice: during and after office hours. If the patient does not answer the phone, the investigators will also send a text message to inform them about the reason for our attempted phone call.

Questionnaire (symptoms and characteristics):

Our multidisciplinary team of clinicians, methodologists, and patient partners developed a questionnaire that records basic patient information. This questionnaire has already been in use with the long-term follow-up of patients who received remdesivir in the SOLIDARITY Finland trial. The questions include i) date of completing the questionnaire, ii) age, iii) height and weight, iv) smoking status (never, ex-smoker, current smoker), v) possible comorbidities, and whether diagnosed before or after COVID-19-infection (obstructive sleep apnea, stroke, coronary artery disease, diabetes, hypertension, cancer, and any psychiatric disease), vi) employment (student, unemployed, employed, sickness allowance, retired), vii) working capability in comparison to the pre-COVID-19 state, viii) physician visits due to symptoms associated with COVID-19, ix) physician-diagnosed long-COVID-19 syndrome. Questionnaires will also document long-term symptoms. Relevant long-COVID-19 -symptoms (in total 20) were identified from recent publications and review articles. This same questionnaire will be used at one and two years. Exertional and cardiopulmonary symptoms potentially related to COVID include fatigue, postexertional malaise, dyspnea during exercise, chest discomfort, palpitations, cough, and respiratory mucous discharges. Main neuropsychiatric symptoms potentially related to COVID include generalized fatigue, attention and memory deficits, sleeping difficulties, depression and anxiety, dizziness, and even sensory disturbances such as paresthesias and changes in taste or smell perceptions. Other commonly encountered symptoms potentially related to COVID include widespread pains (muscle and joint pains, headache), skin rash, nausea, and fever. The burden from each individual symptom is an ordinal variable and will be graded from 0 to 3, where 0 represents no symptom, 1 represents mild bother, 2 moderate bother, and 3 severe bother due to the symptom. Dyspnea is assessed in accordance with the Modified Medical research council dyspnea scale (mMRC) from 0 to 4, where 0 represents dyspnea only with strenuous exercise, and 4 the presence of dyspnea even with mild physical activity, e.g., dressing clothes. To capture the dimensions of recovery, the investigators will use the Core Outcome Measure for Recovery, which has been recommended for use in COVID-19 research.

Quality of life:

The investigators have obtained permission from EuroQol to use the EQ-5D-5L questionnaire to record the patient's QoL. EQ-5D-5L assesses the domains of mobility, self-care, usual daily activities, general pain/discomfort, anxiety/depressions, and an overall impression of health. The first five domains are graded from 1 to 5, while the last uses the visual analogue scale from 0 to 100. Due to our multiethnic patient population, the questionnaires have been translated into the following languages: Albanian, Arabic, English, Estonian, Farsi, Finnish, Russian, Somali, and Swedish. The above-mentioned questionnaire (Finnish language version as the original) has also been translated into these languages.

Data security and future use of data:

Patient information will be encrypted and held securely by the Sponsor. Those analyzing it will use only pseudonymized data, and no identifiable patient details will appear in publications. Data from questionnaires will also be analyzed using pseudonymized data. The investigators have taken care to limit the questions to necessary and clinically relevant aspects related to long COVID.

Primary outcome variables:

i) Symptoms: Each 20 symptoms between the two treatment arms will be compared. These are measured as follows; each range from 0 to 3 (0 = No symptom. 1 = Symptom exists and causes small bother. 2 = Symptom exists and causes moderate bother. 3 = Symptom exists and causes severe bother.) ii) QoL: Using the EQ-5D-5L to compare domain-specific scores between the two treatment arms.

Additional variables (at 1 or 2 years; depending on future funding and ethical approval decisions; currently the study has ethical approval for long-COVID and quality of life assessments only):

* Registry data: Mortality data will be obtained from Digital and Population Data Services Agency (Finnish Digital Agency)). Underlying causes of death will be obtained from Statistics Finland and classified according to the International Statistical Classification of Diseases and Related Health Problems, 10th revision). In line with the Finnish regulations, any consent will not be required from the study patients to acquire information on their census data, vital status, and causes of death for registry research purposes. Comorbidity will be obtained from Finnish Institute for Health and Welfare THL. These will be performed through linkage the patient national identification number to registry records. This study is unlikely well-powered to measure changes in mortality; however, being aware of the vital status is important for the overall follow-up of study participants.
* Spirometry parameters are continuous variables as absolute values (liters = L; liters per second = L/s), percentage of reference values, and z-values. These include VC, FVC, FEV1, FEV1/VC, peak expiratory flow (PEF), the maximal expiratory flow at 50 % (MEF50), and the forced expiratory time (FET). Spirometry will be performed with a bronchodilator test to assess the changes between baseline and after bronchodilation. Diffusing capacity parameter DLCO is a continuous variable with ml/min/mmHg as the unit.
* Entire genomes will be sequenced to identify single-nucleotide polymorphisms that would associate with long-COVID symptoms and the effect of imatinib or infliximab.

Subgroup analyses:

For the primary outcomes, a priori planned subgroup analysis will be performed for whether the patient needed oxygenation at hospital admission (the investigators hypothesize that the treatment effect is larger for those without extra oxygen than those with extra oxygen at hospital admission).

Comparisons between the two treatment arms will be performed as follows:

* Descriptive statistics: Descriptive statistics will be presented with numbers and percentages for categorical variables and means, standard deviation, and range for continuous variables. In the case of clearly skewed continuous variables, they will be presented with median, interquartile range (25th and 75th percentiles), and range. Demographics and baseline characteristics will be presented with descriptive statistics without any hypothesis testing.
* Continuous variables will be subject to repeated measures mixed models or appropriate non-parametric alternatives.
* Binary response variables will be analyzed using logistic regression (possibly adjusting for within-subject dependencies by generalized estimating equations or mixed models) or chi-square/Mantel-Haenszel tests.
* If missing data is regarded as having a significant effect on the conclusions of the trial, sensitivity analyses with different methods for handling missing data will be included.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients, 18 years and above
* SARS-2-CoV-2 infection, laboratory-confirmed
* Admission to the hospital ward or ICU
* Written informed consent prior to initiation of the study or a close relative/legal representative provides written informed consent prior to initiation of the study according to the presumed will of the patient when the patient is unable to give consent herself/himself.
* No anticipated transfer within 72 hours to a non-study hospital

Exclusion Criteria:

* Estimated life expectancy under three months due to severe comorbidity
* ASAT/ALAT-ratio over five-fold upper limit
* Acute myocardial infarction or unstable angina pectoris
* Breast feeding or pregnancy
* Any reason why, in the opinion of the investigators, the patient should not participate
* Patient participates in a potentially confounding drug or device trial during the course of the study
* Already receiving any of the study drugs
* Severe renal failure (eGFR < 30 mL/min)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2022-02-06 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Long-COVID symptoms | At six months from hospital admission.
  Specific questionnaire for symptoms and their severity
Long-COVID symptoms | At one year from hospital admission.
  Specific questionnaire for symptoms and their severity
Long-COVID symptoms | At two years from hospital admission.
  Specific questionnaire for symptoms and their severity
Health-related quality of life | At six months from hospital admission
  EQ-5D-5L questionnaire
Health-related quality of life | At one year from hospital admission
  EQ-5D-5L questionnaire
Health-related quality of life | At two years from hospital admission
  EQ-5D-5L questionnaire

SECONDARY OUTCOMES:
Mortality | During one and two years from hospital admission
  Obtained from health care registries
Incidence of comorbidity | During two years from hospital admission
  Obtained from health care registries
Lung function | At two years from hospital admission
  Spirometry
Lung function | At two years from hospital admission
  Lung diffusion capacity
Lung function | At two years from hospital admission
  6-minute walking test
Whole-genome sequencing | Within 2 years from hospital discharge

CONTACTS AND LOCATIONS:
Overall Officials: Kari AO Tikkinen, MD PhD, Study Director — University of Helsinki
Locations (1):
- University of Helsinki, Helsinki, Finland